CLINICAL TRIAL: NCT05982171
Title: Transcutaneous Spinal Cord Stimulation to Promote Walking Recovery After Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#2023877
Record Dates: First submitted 2023-07-24; First posted 2023-08-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Exoskeleton+Transcutaneous Spinal Cord Stimulation (Experimental): Treatment in this group will involve walking overground using the assistance of an exoskeleton while receiving a therapeutic level of transcutaneous spinal cord stimulation (TSCS) thoracolumbar spinal cord areas. Focus will be on stepping at a high intensity throughout the session as measured by heart rate.
  Interventions: Device: Exo + TSCS
- Exoskeleton+Sham Stimluation (Sham Comparator): Treatment in this group will involve walking overground using the assistance of an exoskeleton while receiving a non-therapeutic level of stimulation (considered to be a sham). Focus will be on stepping at a high intensity throughout the session as measured by heart rate.
  Interventions: Device: Exo + Sham

INTERVENTIONS:
Device: Exo + TSCS — Participants will receive TSCS delivered with the ONWARD Lift system at 1ms using a 10kHz carrier frequency delivered at 30Hz, with an amplitude set for each participant based on their ability to increase voluntary movement output.
  Arms: Exoskeleton+Transcutaneous Spinal Cord Stimulation
Device: Exo + Sham — The ONWARD Lift system will also be used to deliver sham stimulation which will also be delivered at 1ms using a 10kHz carrier frequency delivered at 30Hz, and an amplitude of 1ma which has been used in other sham stimulation protocols and is not sufficient to induce activation of lumbosacral neuronal pools.
  Arms: Exoskeleton+Sham Stimluation

SUMMARY:
The goal of this clinical trial is to investigate the effects of transcutaneous spinal cord stimulation (TSCS) combined with exoskeleton training, as compared to exoskeleton training alone to improve motor function in individuals with incomplete spinal cord injury who are 12 months or less post-injury. Participants will be randomly assigned to a treatment group (exoskeleton training with TSCS, or exoskeleton training without TSCS). Participants in both groups will undergo a baseline evaluation, then take part in 24, 1-hour training sessions at Craig Hospital. After the 24 sessions have concluded, participants will undergo a post-treatment evaluation as well as a follow-up evaluation four weeks after training is completed. Researchers will compare the two groups by evaluating the following areas:

* walking ability and speed
* lower extremity strength, activation, and spasticity
* trunk control
* bowel and bladder function

ELIGIBILITY:
Inclusion Criteria:

* < 12 months post traumatic iSCI C4-T10 with signs of upper motor neuron injury
* AIS C or D classification
* 18 years and older
* Height 5'0" to 6'4"
* Weight 220lbs or less
* Sufficient upper extremity strength to manage a stability aide
* Medical clearance for high intensity gait training
* Walking <1.46 m/s
* Intact skin in on pelvis, lower extremities and back
* Passive range of motion at shoulders, trunk, hips, knees & ankles within functional limits

Exclusion Criteria:

* Unstable or symptomatic cardiac or respiratory issues
* Recent history of fracture, contractures, pressure injury, deep vein thrombosis, or other infection that might interfere with participation in study
* Received Botox injections to the lower extremities within the last six months
* Pregnancy
* Cauda Equina injury
* Any other issue that in the opinion of the investigator would impact study participation
* Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in score on Walking Index for SCI (WISCI) II | Baseline to Immediately After Intervention
  Assesses the amount of physical assistance/devices needed for walking following paralysis from SCI (scale of 0-20 with higher score indicating less need for assistance)

SECONDARY OUTCOMES:
Change in walking speed as measured by the 10 Meter Walk Test | Baseline to Immediately After Intervention
  Participants walk a ten-meter track; time to walk the middle six meters is recorded and converted to meters/second (speed)
Change in distance walked as measured by the 6 Meter Walk Test | Baseline to Immediately After Intervention
  Measures distance walked (in meters) over 6 minute time period
Change in lower extremity strength as measured by Lower Extremity Motor Score (LEMS) | Baseline to Post-treatment
  Assesses strength in 10 lower extremity muscle groups (each muscle scored 0-5 with higher score for greater strength; total score ranges 0-50.
Change in spasm frequency and severity as measured by Penn Spasm Frequency | Baseline to Immediately After Intervention
  Self-report measure of perception of spasticity frequency (0 to 5 scale with higher score more frequent spasms) and severity (1-3 scale with higher score more severe spasms)
Change in bowel function as measured by Neurogenic Bowel Dysfunction Scale | Baseline to Immediately After Intervention
  Symptom based questionnaire evaluating bowel dysfuntion and its impact on quality of life (score 0-47 with higher score indicating greater bowel dysfunction)
Change in bladder function as measured by Neurogenic Bladder Symptom Scale | Baseline to Immediately After Intervention
  Symptom based questionnaire evaluating bladder function and its impact on quality of lifehe Neurogenic Bladder Symptom Score (NBSS) is a validated 24 item questionnaire that measures bladder symptoms across 3 different domains: incontinence (scored 0-29), storage and voiding (scored 0-22), and consequences (scored 0-23); there is a single general urinary QOL question scored from 0 (pleased) to 4 (unhappy
Change in balance/trunk control as measure by the Function in Sitting Test Spinal Cord Injury | Baseline to Immediately After Intervention
  Assesses static, proactive, and reactive balance as well as sensory integration. Each area assessed on scale of 0-4 with higher score indicating more independent trunk control.

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No